CLINICAL TRIAL: NCT06354998
Title: Randomized, Observer-Blind, Active-Controlled, Clinical Trial to Assess the Immunogenicity of an Investigational mRNA-1273.815 COVID-19 Vaccine in Previously Vaccinated Adults
Brief Title: A Study of an Investigational mRNA-1273.815 COVID-19 Vaccine in Previously Vaccinated Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P401
Record Dates: First submitted 2024-04-05; First posted 2024-04-09 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273.815; mRNA-1273.815 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Investigational mRNA-1273.815 (Experimental): Participants will receive Investigational mRNA-1273.815 by intramuscular injection.
  Interventions: Biological: Investigational mRNA-1273.815
- Licensed Spikevax Vaccine (Active Comparator): Participants will receive a licensed Spikevax vaccine by intramuscular injection.
  Interventions: Biological: Licensed Spikevax Vaccine

INTERVENTIONS:
Biological: Investigational mRNA-1273.815 — Sterile solution for injection
  Arms: Investigational mRNA-1273.815
Biological: Licensed Spikevax Vaccine — Commercially available formulation
  Arms: Licensed Spikevax Vaccine

SUMMARY:
To evaluate immune responses of an Investigational mRNA-1273.815 vaccine against the Omicron subvariant strain (XBB.1.5) of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

ELIGIBILITY:
Inclusion Criteria:

* Participants of childbearing potential may be enrolled in the study if the participant fulfills all of the following criteria:

  1. Has a negative pregnancy test on the day of injection prior to vaccine dose being administered (Day 1).
  2. Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1.
  3. Has agreed to continue using an effective contraception through 2 weeks following injection.
  4. Is not currently breastfeeding.

Exclusion Criteria:

* Has known history of SARS-CoV-2 infection within 3 months prior to enrollment.
* Currently has symptomatic acute or unstable chronic disease requiring medical or surgical care, to include significant change in therapy or hospitalization for worsening disease, at the discretion of the Investigator.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the Investigator's judgment.
* Reported history of congenital or acquired immunodeficiency (for example, human immunodeficiency virus), immunosuppressive condition, asplenia, or recurrent severe infections disease.
* Has known or suspected allergy or history of anaphylaxis, urticaria, or other significant adverse reaction to the vaccine or its excipients.
* Receipt of the following:

  1. COVID-19 vaccine within 3 months prior to enrollment
  2. Any other licensed vaccine within 28 days before or 2 weeks after the study injection, with the exception of influenza vaccines, which may be given 14 days before or after receipt of a study vaccine.
  3. Systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥10 milligrams/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study. Note: Inhaled, nasal, and topical steroids are allowed.
  4. Systemic immunoglobulins or blood products within 3 months prior to Screening or plans for receipt during the study.
* Has donated ≥450 milliliters of blood products within 28 days prior to Screening or plans to donate blood products during the study.
* Has participated in an interventional clinical study within 28 days prior to Screening or plans to participate in an interventional clinical trial of an investigational vaccine or drug while participating in this study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Paratus Canberra, Canberra, Australian Capital Territory
  - Holdsworth House, Darlinghurst, New South Wales
  - Paratus Brisbane, Brisbane, Queensland
  - USC Morayfield, Morayfield, Queensland
  - University of the Sunshine Coast, South Bank, South Brisbane, Queensland
  - Emeritus Melbourne, Camberwell, Victoria
  - AusTrials Sunshine Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational mRNA-1273.815: Participants received Investigational mRNA-1273.815 by intramuscular (IM) injection on Day 1.
- Licensed Spikevax Vaccine: Participants received a licensed Spikevax vaccine by IM injection on Day 1.
Period: Overall Study
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine
Started | 108 | 109
Received Study Vaccination | 106 | 109
Completed | 105 | 109
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all enrolled participants who received study drug.
Groups:
- Investigational mRNA-1273.815: Participants received Investigational mRNA-1273.815 by IM injection on Day 1.
- Total: Total of all reporting groups
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine | Total
Number analyzed (Participants) | 106 | 109 | 215
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (16.09) | 46.0 (17.47) | 47.1 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 58 | 57 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 93 | 85 | 178
  Unknown or Not Reported | 10 | 19 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 82 | 92 | 174
  Race: Black or African American | 1 | 1 | 2
  Race: Asian | 12 | 10 | 22
  Race: Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  Race: Multiple | 2 | 3 | 5
  Race: Other | 7 | 2 | 9
  Race: Not reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean (GM) Value of Neutralizing Antibodies (nAbs) Against SARS-CoV-2-specific Strain at Day 15
Description: Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5 * LLOQ. Values reported greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ if actual values were not available. LLOQ was 38 arbitrary unit (AU)/milliliter (mL) and ULOQ was 6960 AU/mL. 95% confidence interval (CI) of GM value was calculated based on the t-distribution of the log-transformed values for antibodies, then back transformed to the original scale for presentation.
Time Frame: Day 15
Population: The Per-protocol Immunogenicity Subset (PPIS) included participants who received planned dose of study injection per schedule, complied with immunogenicity testing schedule and had no major protocol deviations that impacted key or critical data.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine
Number analyzed (Participants) | 103 | 104
AU/mL | 1180.55 [927.67 to 1502.38] | 1300.25 [1056.39 to 1600.40]
Statistical Analysis 1: Comparison: Investigational mRNA-1273.815 vs Licensed Spikevax Vaccine; GMR (mRNA-1273.815 versus licensed Spikevax) at Day 15 and its 95% CI was calculated based on the t-distribution for the mean difference of log-transformed antibody values and then back transformed to the original scale for presentation; Test type: Other; Geometric Mean Ratio (GMR) = 0.908, 95% CI 2-sided [0.662 to 1.245] — GMR was a secondary endpoint

2. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) of Special Interest (AESIs), and AEs Leading to Withdrawal From the Study
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. Number of participants with SAEs, AESIs, and AEs leading to discontinuation up to Day 15 are reported in this outcome measure. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 15
Population: Safety Set included all enrolled participants who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine
Number analyzed (Participants) | 106 | 109
Participants
  SAEs | 1 | 0
  AESIs | 0 | 0
  AEs Leading to Withdrawal | 0 | 0

3. Secondary Outcome: Seroresponse Rate of nAb Against the SARS-CoV-2-specific Strain: Percentage of Participants With Seroresponse
Description: Seroresponse at a participant level was defined as a change from baseline below the LLOQ to equal or above 4 * LLOQ, or at least a 4-fold rise if baseline was equal to or above the LLOQ. LLOQ was 38 AU/mL.
Time Frame: Day 15
Population: The PPIS included participants who received planned dose of study injection per schedule, complied with immunogenicity testing schedule and had no major protocol deviations that impacted key or critical data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine
Number analyzed (Participants) | 103 | 104
percentage of participants | 66.0 [56.0 to 75.1] | 69.2 [59.4 to 77.9]

ADVERSE EVENTS:
Time Frame: Day 1 through Day 15
Description: The all-cause mortality was based on the randomization set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all enrolled participants who received the study drug.
Arm/Group | Investigational mRNA-1273.815 | Licensed Spikevax Vaccine
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/109
Serious Adverse Events (participants affected / at risk) | 1/106 | 0/109
Other Adverse Events (participants affected / at risk) | 0/106 | 0/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational mRNA-1273.815 (N=106) | Licensed Spikevax Vaccine (N=109)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT06354998/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT06354998/SAP_001.pdf